CLINICAL TRIAL: NCT02536092
Title: A Prospective Multi-Center Study of a Novel Dual-Wavelength Laser for Hair Removal
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor terminated study
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-15-HR-03
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Hypertrichosis
MeSH Terms: conditions — Hypertrichosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 755nm and 1064nm Nd:YAG laser (Experimental): 755nm and 1064nm Nd:YAG laser
  Interventions: Device: 755nm and 1064nm Nd:YAG laser

INTERVENTIONS:
Device: 755nm and 1064nm Nd:YAG laser — Dual wavelength 755nm and 1064nm Nd:YAG laser
  Other Names: Excel HR

SUMMARY:
To evaluate the safety and efficacy of the Cutera excel HR dual wavelength 755nm Alexandrite and 1064nm Nd:YAG laser for hair removal.

DETAILED DESCRIPTION:
This is a multi-center prospective, open-label, uncontrolled multi-center study of up to 50 male or female subjects, age 18 to 65 years, who desire laser hair removal. Subjects will receive 6 hair removal treatments, spaced 8 weeks apart, and will be followed at 12 weeks post-final treatment.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male, 18 to 65 years of age (inclusive).
* Fitzpatrick Skin Type I - VI (Appendix 3).
* Subject has black or dark brown unwanted hair.
* Subject must be able to read, understand and sign the Informed Consent Form.
* Must be willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions.
* Willing to refrain from shaving the treatment area for 5 days prior to each study visit.
* Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, educational or marketing purposes.
* Must agree not to use hair removal products, such as topical chemical depilatories, or undergo any other hair removal procedure during the study, such as other laser and light therapies or waxing.
* Willing to refrain from excess sun exposure and willing to wear sunscreen on the treatment area during the study (including the follow-up period).
* Be in good health, as determined by the Investigator.
* Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study

Exclusion Criteria:

* Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
* Had any type of professional hair removal procedure, such as laser, light-based, RF or electrolysis, in the treatment area within 12 months of study participation.
* Had other epilation treatment, such as waxing or mechanical epilator, in the treatment area within 6 months of study participation.
* Subject shows signs of actinic bronzing or recent tanning in the treatment area, and unable/unlikely to refrain from tanning during the study
* History of malignant tumors in the target area.
* Pregnant and/or breastfeeding.
* Having an infection, dermatitis or a rash in the treatment area.
* Significant concurrent illness, such as diabetes mellitus or cardiovascular disease, e.g., uncontrolled hypertension.
* Suffering from coagulation disorders or taking prescription anticoagulation medications.
* History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
* Currently using immunosuppressive medications or history of immunosuppression/immune deficiency disorder, such as psoriasis, eczema, vitiligo, systemic lupus erythematosus or scleroderma.
* History of seizure disorders due to light.
* Any use of medication that is known to increase sensitivity to light according to Investigator's discretion.
* History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen
* History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
* History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation.
* Systemic use of corticosteroid or isotretinoin within 6 months of study participation.
* Anytime in life, having have used gold therapy (gold salts) for disorders such as rheumatologic disease or lupus.
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study.
* Current smoker or history of smoking within 6 months of study participation.
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Physician's Global Assessment | 12 weeks
  Percentage of hair reduction

SECONDARY OUTCOMES:
Incidence and severity of adverse device effects | 12 weeks
  Assessment of ADEs immediately following each laser treatment and at the final follow-up visit

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Lezara Laser & Vein Care, Squamish, British Columbia
  - Body Bar Laser Clinic/Academy, Surrey, British Columbia

IPD SHARING:
Plan to Share IPD: No
Study terminated